CLINICAL TRIAL: NCT07138989
Title: Efficacy and Safety of EBV Lytic Reactivation Therapy Combined With PD-1 Antibody in Recurrent/Metastatic Nasopharyngeal Carcinoma: a Single-center, Single-arm Phase II Trial
Brief Title: EBV Lytic Reactivation Therapy Combined With PD-1 Antibody in Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-184
Record Dates: First submitted 2025-08-11; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; Epstein-Barr virus; immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — Valganciclovir; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- EBV Lytic Reactivation Therapy (Experimental): Patients will receive 4 to 6 cycles of gemcitabine, cisplatin, and PD-1 antibody, with oral administration of valganciclovir hydrochloride tablets during the first 3 cycles. Following completion of 4 to 6 cycles, patients will continue with maintenance therapy using PD-1 antibody.
  Interventions: Drug: Valganciclovir Hydrochloride Tablets; Drug: gemcitabine, cisplatin, and PD-1 antibody

INTERVENTIONS:
Drug: Valganciclovir Hydrochloride Tablets — Valganciclovir hydrochloride tablets will be administered at 900 mg twice daily from day 1 to day 14, followed by 450 mg twice daily from day 15 to day 20, for a total of 3 cycles.
Drug: gemcitabine, cisplatin, and PD-1 antibody — Gemcitabine 1000 mg/m² will be administered intravenously on days 1 and 8; cisplatin 80 mg/m² intravenously on day 1; and PD-1 antibody intravenously on day 1. Each cycle is 21 days in duration, and treatment will be administered for a total of 4 to 6 cycles.
  Following completion of the 4 to 6 cycles, patients will continue PD-1 antibody maintenance therapy (every 3 weeks) for up to two years or until disease progression, unacceptable toxicity, initiation of a new anticancer therapy, withdrawal of informed consent, or death.

SUMMARY:
Nearly all undifferentiated nasopharyngeal carcinoma (NPC) are associated with the Epstein-Barr Virus (EBV), which typically remains in a latent, non-immunogenic state within tumor cells. By combining EBV lytic induction strategy with standard chemo-immunotherapy, this study aims to create a synergistic anti-tumor effect and improve clinical outcomes for patients with recurrent/metastatic NPC (r/m NPC). This is a phase II, single-center, single-arm clinical trial designed to evaluate the efficacy and safety of a novel combination therapy in patients with r/m EBV-positive NPC.

DETAILED DESCRIPTION:
Rationale: Epstein-Barr virus (EBV) is clonally present in nearly all undifferentiated nasopharyngeal carcinoma (NPC) tumor cells, particularly in endemic regions. In most cases, EBV remains in a latent state, expressing only a limited set of non-immunogenic proteins, which facilitates immune evasion by tumor cells. Chemotherapeutic agents such as gemcitabine and cisplatin can induce the EBV lytic cycle, activate valganciclovir hydrochloride, thereby enabling the selective killing of EBV-infected tumor cells. This strategy may act synergistically with immunotherapy. Early-phase clinical studies have demonstrated the safety and potential efficacy of this approach; however, larger-scale studies are required to confirm these findings.

Study Objectives: The primary objectives of this clinical trial are: 1.To assess the objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), duration of response (DoR), and overall survival (OS) in patients receiving chemotherapy combined with valganciclovir hydrochloride and PD-1 antibody. 2.To evaluate the safety profile, including acute and chronic toxicities.

Study Design and Treatment Regimen: Patients with histologically confirmed EBV-positive, recurrent or metastatic NPC will be enrolled. Patients will receive 4 to 6 cycles of gemcitabine, cisplatin, and PD-1 antibody, with oral administration of valganciclovir hydrochloride tablets during the first 3 cycles. Following completion of the 4 to 6 cycles, patients will continue PD-1 antibody maintenance therapy for up to two years or until disease progression, unacceptable toxicity, initiation of a new anticancer therapy, withdrawal of informed consent, or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must voluntarily participate and provide written informed consent.
* Histologically or cytologically confirmed recurrent or metastatic nasopharyngeal carcinoma (NPC) at enrollment, with positive EBERs by pathological immunohistochemistry.
* Metastatic NPC includes both newly diagnosed metastatic disease and metastatic disease after failure of first-line therapy, as well as recurrent NPC not amenable to local regional treatment, with confirmed metastatic or recurrent disease and no prior treatment after diagnosis.
* Age ≥ 18 years and ≤ 75 years, of any sex.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival time ≥ 3 months.
* Baseline plasma EBV DNA > 0 copies/mL.
* Adequate organ function confirmed by the following criteria (no blood component transfusions or use of hematopoietic growth factors within 2 weeks prior to study treatment initiation):
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet count ≥ 100 × 10^9/L; hemoglobin ≥ 90 g/L. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or calculated creatinine clearance (CrCl) ≥ 60 mL/min . Total bilirubin (TBil) ≤ 1.5 × ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (for patients with liver metastases, TBil ≤ 3 × ULN; AST and ALT ≤ 5 × ULN). Serum albumin ≥ 28 g/L.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other monoclonal antibodies or to any component of PD-1 inhibitors.
* Receipt of radiotherapy, biological therapy (e.g., tumor vaccines, cytokines, or growth factors), or other immunotherapy (excluding PD-1 and PD-L1 inhibitors), or any other anti-tumor treatment within 28 days or 5 half-lives prior to the first dose of study drug, whichever is shorter.
* Prior treatment targeting Epstein-Barr virus (EBV) specifically.
* History of any Grade ≥3 bleeding event, as defined by CTCAE v5.0, within 4 weeks prior to screening, or patients deemed at high risk of bleeding by the investigator.
* Presence of necrotic lesions within 4 weeks prior to screening, with high risk of major hemorrhage as judged by the investigator.
* Known congenital or acquired immunodeficiency (e.g., HIV-positive individuals).
* Requirement for systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive agents within 14 days prior to initiation of study treatment.
* History of active tuberculosis (TB). Suspected active TB must be excluded through chest X-ray, sputum examination, and clinical assessment of signs and symptoms.
* Patients with HBV DNA ≥1000 copies/mL. Patients with positive hepatitis C antibody results may only be enrolled if polymerase chain reaction (PCR) testing confirms HCV RNA negativity.
* Pregnant or breastfeeding women, or women of childbearing potential not using effective contraception.
* History of other malignancies, except for adequately treated basal cell carcinoma or carcinoma in situ of the cervix.
* Uncontrolled cardiovascular conditions, including but not limited to: Heart failure with NYHA classification ≥2; Unstable angina; Myocardial infarction within the past year; Supraventricular or ventricular arrhythmias requiring treatment or intervention.
* Significant impairment of cardiac, hepatic, pulmonary, renal, or bone marrow function.
* Severe and uncontrolled medical illnesses or infections.
* Concurrent participation in another clinical trial or use of another investigational agent.
* Refusal or inability to sign informed consent.
* Any other contraindications to study treatment as determined by the investigator.
* Individuals with personality disorders or psychiatric conditions, and those lacking or having limited legal capacity to provide consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-19 (Estimated); Primary Completion 2026-08-18 (Estimated); Study Completion 2031-08-18 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | From enrollment to the end of treatment. Up to 2 approximately years.
  Objective Response Rate (ORR) is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 from the National Cancer Institute (NCI).

SECONDARY OUTCOMES:
Disease Control Rate，DCR | From enrollment to the end of treatment. Up to 2 approximately years.
  Disease Control Rate (DCR) is defined as the proportion of patients who achieve tumor response classified as partial response (PR), complete response (CR), or stable disease (SD) according to recognized response evaluation criteria-such as RECIST version 1.1.
Progression-free Survival, PFS | 1 years; 2 years; 5 years;
  Defined as the time from registration to documented disease progression or non-cancer-specific death.
Duration of Response, DoR | From enrollment to disease progression. Up to 2 approximately years.
  Defined as the median length of time from the initial documentation of a tumor response (either complete response [CR] or partial response [PR]) to disease progression or death from any cause.
Overall Survival, OS | 1 years; 2 years; 5 years
  Defined as the time from registration to death from any cause.
Incidence rate of acute and late adverse events (AEs) | From enrollment to the end of follow-ups. Up to 2 approximately years.
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Qiang Mai, MD,PhD, Principal Investigator — Sun Yat-sen Universitty Cancer Center
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted to the Research Data Deposit (RDD) public platform (http://www.researchdata.org.cn) and available from the principal investigators upon reasonable request.

REFERENCES:
- [Background] Ghosh SK, Perrine SP, Williams RM, Faller DV. Histone deacetylase inhibitors are potent inducers of gene expression in latent EBV and sensitize lymphoma cells to nucleoside antiviral agents. Blood. 2012 Jan 26;119(4):1008-17. doi: 10.1182/blood-2011-06-362434. Epub 2011 Dec 7. PMID 22160379
- [Background] Perrine SP, Hermine O, Small T, Suarez F, O'Reilly R, Boulad F, Fingeroth J, Askin M, Levy A, Mentzer SJ, Di Nicola M, Gianni AM, Klein C, Horwitz S, Faller DV. A phase 1/2 trial of arginine butyrate and ganciclovir in patients with Epstein-Barr virus-associated lymphoid malignancies. Blood. 2007 Mar 15;109(6):2571-8. doi: 10.1182/blood-2006-01-024703. Epub 2006 Nov 21. PMID 17119113
- [Background] Wu M, Hau PM, Li L, Tsang CM, Yang Y, Taghbalout A, Chung GT, Hui SY, Tang WC, Jillette N, Zhu JJ, Lee HHY, Kong EL, Chan MSA, Chan JYK, Ma BBY, Chen MR, Lee C, To KF, Cheng AW, Lo KW. Synthetic BZLF1-targeted transcriptional activator for efficient lytic induction therapy against EBV-associated epithelial cancers. Nat Commun. 2024 May 3;15(1):3729. doi: 10.1038/s41467-024-48031-8. PMID 38702330
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi Y, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Wang S, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Luo X, Wang X, Tang X, Feng H, Yao S, Keegan P, Xu RH. Toripalimab Plus Chemotherapy for Recurrent or Metastatic Nasopharyngeal Carcinoma: The JUPITER-02 Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1961-1970. doi: 10.1001/jama.2023.20181. PMID 38015220